CLINICAL TRIAL: NCT02055222
Title: Clinical Outcomes and Molecular Phenotypes in Smokers With Parenchymal Lung Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140049; 14-H-0049
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Fibrosis; Lung Disease
Keywords: COPD; Smoking; Idiopathic Pulmonary Fibrosis; Natural History
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases; Pulmonary Disease, Chronic Obstructive; Smoking; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lung disease (IPF) and smoking history: 50 IPF and 50 COPD patients, and 30 subjects with early interstitial lung abnormalities seen on previous radiographs
- Lung disease COPD and smoking history: 50 IPF and 50 COPD patients, and 30 subjects with early interstitial lung abnormalities seen on previous radiographs
- Normal Volunteers- Non-smokers, and Smokers: 50 smoking and 30 non-smoking controls

SUMMARY:
Despite the implementation of modern public health interventions, 1 in 5 adults in the United States are either current or former smokers and remain at risk for the development of chronic lung diseases. It is unknown how or why any one individual smoker can develop a wide range of lung diseases including chronic obstructive lung disease and/or pulmonary fibrosis. The purpose of this protocol is to collect clinical data, blood, urine, and bronchoalveolar samples from smokers and non-smokers in an attempt to establish phenotypic clinical profiles that correspond to divergent pathways in the expression of such proteins as the transforming growth factor-beta1 (TGF-beta <=1). The information generated from this study will provide insight into the pathogenesis of smoking-related lung injury and potentially allow for the development of early therapeutic interventions.

DETAILED DESCRIPTION:
Despite the implementation of modern public health interventions, 1 in 5 adults in the United States are either current or former smokers and remain at risk for the development of chronic lung diseases. It is unknown how or why any one individual smoker can develop a wide range of lung diseases including chronic obstructive lung disease and/or pulmonary fibrosis. The purpose of this protocol is to collect clinical data, blood, urine, and bronchoalveolar samples from smokers and non-smokers in an attempt to establish phenotypic clinical profiles that correspond to divergent pathways in the expression of such proteins as the transforming growth factor-beta1 (TGF-beta1). The information generated from this study will provide insight into the pathogenesis of smoking-related lung injury and potentially allow for the development of early therapeutic interventions.

ELIGIBILITY:
* INCLUSION CRITERIA: For subjects with lung diseases:
* Men and women age 40-80 years
* Smokers with greater than or equal to 10 pack-year history of ever-smoking

EXCLUSION CRITERIA: For subjects with lung diseases:

Subjects will be excluded from the study if they meet one or more of the following criteria:

* Subjects who are under the age of 40 or over 80 years old
* Women who are pregnant or lactating
* Have known allergies to lidocaine or medications used for moderate sedation
* Active coronary artery disease
* Cerebral-vascular accident within the past 12 months
* Active anticoagulation
* Active infections
* Cancer, or a history of cancer within the previous 5 years of screening (other than adequately treated cutaneous basal cell, squamous cell carcinoma, excised melanoma, or carcinoma in situ of the uterine cervix with no evidence of recurrence).
* Poorly controlled chronic diseases
* Unable to provide consent
* Impaired renal function (including dialysis)
* Contraindications to MRI scan including:

  * electrical implants such as cardiac pacemakers or perfusion pumps
  * ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
  * ferromagnetic objects such as jewelry or metal clips in clothing
  * pre-existing medical conditions, including a likelihood of developing seizures or anxiety disorders such as claustrophobia, panic attacks or any psychiatric disorder

INCLUSION CRITERIA: For Non-Smoking Controls

* Men and women age 40-80 years
* No prior history of smoking (this is a non-smoking cohort)

EXCLUSION CRITERIA: For Non-Smoking Controls

* Subjects who are under the age of 40 or over 80 years old
* Women who are pregnant or lactating
* Have known allergies to lidocaine or medications used for moderate sedation
* Active coronary artery disease
* Cerebral-vascular accident within the past 12 months
* Active anticoagulation
* Active infections
* Cancer, or a history of cancer within the previous 5 years of screening (other than adequately treated cutaneous basal cell, squamous cell carcinoma, excised melanoma, or carcinoma in situ of the uterine cervix with no evidence of recurrence).
* Poorly controlled chronic diseases
* Unable to provide consent
* Impaired renal function (including dialysis)
* Contraindications to MRI scan including:

  * electrical implants such as cardiac pacemakers or perfusion pumps
  * ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
  * ferromagnetic objects such as jewelry or metal clips in clothing
  * pre-existing medical conditions, including a likelihood of developing seizures or anxiety disorders such as claustrophobia, panic attacks or any psychiatric disorder

INCLUSION CRITERIA

For Smoking Controls

* Men and women age 40-80 years
* Subjects who have a prior smoking history

EXCLUSION CRITERIA

For Smoking Controls

* Subjects who are under the age of 40 or over 80 years old
* Women who are pregnant or lactating
* Have known allergies to lidocaine or medications used for moderate sedation
* Active coronary artery disease
* Cerebral-vascular accident within the past 12 months
* Active anticoagulation
* Active infections
* Cancer, or a history of cancer within the previous 5 years of screening (other than adequately treated cutaneous basal cell, squamous cell carcinoma, excised melanoma, or carcinoma in situ of the uterine cervix with no evidence of recurrence).
* Poorly controlled chronic diseases
* Unable to provide consent
* Impaired renal function (including dialysis)
* Contraindications to MRI scan including:

  * electrical implants such as cardiac pacemakers or perfusion pumps
  * ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
  * ferromagnetic objects such as jewelry or metal clips in clothing
  * pre-existing medical conditions, including a likelihood of developing seizures or anxiety disorders such as claustrophobia, panic attacks or any psychiatric disorder

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred thirty-eight study subjects with chronic obstructive pulmonary diseases (COPD) and interstitial lung diseases such as idiopathic pulmonary fibrosis (IPF) along with 85 control subjects will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Determine changes in validated clinical parameters of smokers with interstitial lung abnormalities (ILA) as compared to controls and patients with IPF and COPD. | 3 years
  Determine changes in validated clinical parameters of smokers with interstitial lung abnormalities (ILA) as compared to controls and patients with IPF and COPD

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-H-0049.html